CLINICAL TRIAL: NCT07356570
Title: Second Prospective Cohort of Patients Entering the Multidisciplinary Care Pathway for Post-Covid Syndromes - SyPoCo2 Cohort
Acronym: SYPOCO 2
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0943; IDRCB (Other: 2024-A02110-47)
Record Dates: First submitted 2025-06-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: Long COVID; SARS-CoV-2; Post-COVID syndrome; Immune response; Biomarkers; Prospective cohort
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples (30 mL total per patient) will be collected during the inclusion visit: 2 SST tubes (5 mL) and 2 EDTA tubes (10 mL). Samples will be processed for immunological and molecular analyses at Inserm U1111 (CIRI, Lyon) and Inserm We-Met (I2MC, Toulouse).
  All samples will be pseudonymized. No biological specimens will be stored or banked after analysis. DNA and RNA will not be used to identify or re-identify participants.
  No biobank or collection is created as part of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-COVID Patient Cohort: Patients aged ≥18 years with documented SARS-CoV-2 infection and persistent or complex symptoms beyond 4 weeks or 3 months. Participants are referred to either the post-COVID rehabilitation program at Hôpital Henry Gabrielle or the EPSILON pathway at Hôpital Lyon Sud. Clinical and biological data are collected at a single inclusion visit.
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — A one-time 30 mL blood draw is performed during the inclusion visit for immunological and molecular analysis as part of the HERVCOV research program. No therapeutic intervention is administered, and no samples are stored after analysis.

SUMMARY:
The study aims to identify clinical profiles of long-COVID patients and correlate them with immunological and molecular data in order to identify prognostic biomarkers and potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Documented SARS-CoV-2 infection
* Persistent or complex post-COVID symptoms lasting more than 4 weeks or more than 3 months
* Patient referred to the EPSILON pathway or to the post-COVID rehabilitation unit
* Age ≥ 18 years
* Non-institutionalized
* Expected survival greater than 6 months

Exclusion Criteria:

* Refusal to participate or to share data
* Uncontrolled comorbidities
* Pregnant or breastfeeding women
* Persons under legal protection or deprived of liberty
* Not affiliated with the French national health insurance system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: his study involves adult patients (≥18 years) with documented SARS-CoV-2 infection referred to a multidisciplinary post-COVID care pathway. Participants present persistent or complex symptoms beyond 4 weeks or 3 months. Recruitment occurs at Hôpital Henry Gabrielle (rehabilitation unit) and Hôpital Lyon Sud (pulmonology department). Patients are enrolled during their regular clinical follow-up. Clinical and biological data are collected at a single inclusion visit.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants per clinical cluster at Day 0 (clusters derived from unsupervised multivariate analysis of clinical and paraclinical variables). | At inclusion (Day 0), single time point
  At inclusion (Day 0), participants' clinical and paraclinical data will be collected and standardized (z-scores) to derive clinical clusters using unsupervised multivariate methods (principal component analysis for dimensionality reduction if needed, followed by k-means or hierarchical clustering with Euclidean distance).

SECONDARY OUTCOMES:
Differences in clinical and biological parameters between patient subgroups defined by symptom profile and time since initial infection | At inclusion (Day 0)
  atients will be classified into subgroups according to the predominant type and severity of post-COVID symptoms (e.g., fatigue-dominant, cognitive, respiratory) and the interval since acute SARS-CoV-2 infection (<12 months, ≥12 months). Comparative analyses will assess differences in clinical scores (e.g., fatigue, quality of life), and biological markers (e.g., inflammatory cytokines, immune cell subsets) between groups.
Concentration of residual SARS-CoV-2 viral proteins detected in plasma samples at inclusion | At inclusion (Day 0)
  Proteomic analyses (e.g., mass spectrometry, immunoassay) will be performed on plasma samples to quantify the presence of SARS-CoV-2 structural or non-structural proteins (e.g., spike, nucleocapsid).
Serum biomarker concentrations at Day 0 by clinical cluster | Day 0
  Blood is collected at inclusion (Day 0). Each analyte concentration (pg/mL or ng/mL, as applicable) will be summarized per cluster as mean (SD) or median (IQR) and compared across clusters using ANOVA or Kruskal-Wallis with post-hoc tests as appropriate; effect sizes and 95% CIs will be reported.
Association between clinical clusters and serum biomarker panel at Day 0 (standardized mean differences and multivariable models) | Day 0
  Cluster membership will be the exposure; each biomarker (standardized) will be the outcome in linear models adjusted for prespecified covariates (e.g., age, sex, time since first SARS-CoV-2 infection). the investigators will report adjusted differences (β) with 95% CIs and p-values; multiplicity will be handled

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service Pneumologie aigue spécialisée et cancérologie thoracique, Pierre-Bénite
  - Hôpital Henry Gabrielle-HCL, Saint-Genis-Laval

IPD SHARING:
Plan to Share IPD: Undecided